CLINICAL TRIAL: NCT05947838
Title: A Prospective Feasibility Study Using ctDNA to Tailor Neoadjuvant Chemotherapy for Patients With Colorectal or Appendiceal Adenocarcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0214; NCI-2023-05381 (Other: NCI-Clinical Trials Registry)
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Appendiceal Adenocarcinoma; Colorectal
MeSH Terms: conditions — Adenocarcinoma, Mucinous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Circulating tumoral DNA directed neoadjuvant therapy arm (Experimental): Participants will have their circulating tumoral DNA levels measured at the onset of neoadjuvant chemotherapy and during their neoadjuvant treatment to direct the duration of therapy provided.
  Interventions: Procedure: Circulating tumoral DNA directed neoadjuvant therapy arm

INTERVENTIONS:
Procedure: Circulating tumoral DNA directed neoadjuvant therapy arm — Given by IV (vein)

SUMMARY:
To learn if circulating tumor DNA (ctDNA) testing before cytoreductive surgery (CRS) with or without heated intraperitoneal chemotherapy (HIPEC) can show if patients have a low or high risk of the disease returning and help doctors decide if less or more intense chemotherapy is needed as treatment before surgery. ctDNA testing measures the amount of tumor DNA (genetic information) in the blood.

DETAILED DESCRIPTION:
Primary Objectives:

• The primary aim of this prospective study is to assess and compare the recurrence-free survival following CRS and HIPEC of carcinomatosis of colorectal or appendiceal origin with curative intent among ctDNA-negative and ctDNA-positive patients based on their ctDNA status immediately prior to CRS and HIPEC

Secondary Objectives:

* To assess 1 and 2-year recurrence-free survival following CRS and HIPEC with curative intent among ctDNA-negative and ctDNA-positive patients
* To assess and compare 2-year overall survival following CRS and HIPEC among ctDNA-negative and ctDNA-positive patients
* To assess the duration of response, including duration of overall response, duration of overall CR and duration of stable disease
* To evaluate the proportion of ctDNA-negative patients at 1-year post-resection
* To compare survival rate of ctDNA-negative patients undergoing ctDNA-guided postoperative chemotherapy to historical controls
* To evaluate proportion of patients in each arm who change chemotherapy in response to ctDNA measurement
* To delineate the pattern of disease recurrence
* To assess ctDNA sensitivity and specificity for predicting disease recurrence
* To evaluate and correlate patient molecular subtypes and characterization of tumor biologic factors that are associated with ctDNA detection
* To evaluate and correlate cross-sectional imaging characteristics of tumors with biologic factors such as pathologic response, ctDNA detection, and recurrence free survival

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed diagnosis of moderate or poorly differentiated appendiceal or colorectal adenocarcinoma of any grade with Initial resectable disease.
* Have metastatic peritoneal disease that is visible on imaging or at the time of laparoscopy.
* Age ≥18 years. Because no adverse event data are currently available on the use of ctDNA in chemotherapy decision making in patients <18 years of age, children are excluded from this study.
* ECOG performance status ≤1 (Karnofsky ≥70%,).
* Patients must have adequate organ and marrow function as defined below:

absolute neutrophil count ≥1,000/mcL platelets ≥100,000/mcL total bilirubin 1.5x ≤ institutional upper limit of normal (ULN) AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN Creatinine clearance ≥30 mL/min

* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with treated brain metastases are not eligible.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Estimated life-expectancy of > 4 months.
* The effects of standard chemotherapeutic agents used in this trial (5-fluouracil, oxaliplatin, leucovorin, and irinotecan) on the developing human fetus are detrimental. For this reason and because these agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

  * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
  * History of hysterectomy or bilateral salpingo-oophorectomy.
  * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
  * History of bilateral tubal ligation or another surgical sterilization procedure.
* Approved methods of birth control are as follows: Hormonal contraception (i.e., birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of their chemotherapy administration.
* Ability to understand and the willingness to sign a written informed consent document.
* English and Non-English-speaking.

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* Patients who are receiving any other investigational agents.
* Patients with brain or other visceral (i.e. liver and/or lung) metastases at the discretion of the investigator.
* Patients with uncontrolled intercurrent illness (Indicate clearly what type or extent)
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because chemotherapeutic agents used carry the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with chemotherapy, breastfeeding should be discontinued if the mother is treated with chemotherapy. These potential risks may also apply to other agents used in this study.
* If participant received major surgery within last 4 weeks, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
* Serious adverse chemotherapy related adverse events (grade 3 or 4) that were symptomatic and required prolong chemotherapy break (>6weeks).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the study subject's best interest to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
). Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Michael White, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org